CLINICAL TRIAL: NCT04618185
Title: Gut Imaging for Function & Transit in CF - GIFT-CF 3: Evaluation of Triple Combination Therapy.
Brief Title: Gut Imaging for Function & Transit in CF - GIFT-CF 3
Acronym: GIFT-CF3
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Manchester Metropolitan University (Other); Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 20CS036
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
Keywords: Magnetic Resonance Imaging; Oro-caecal transit time; Small bowel water; Colonic volume; Gastrointestinal symptoms; Stool and sputum microbiome; CFTR modulator
MeSH Terms: conditions — Cystic Fibrosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and sputum samples frozen pre-analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- p.Phe508del homozygous genotype: People with CF with 2 copies of p.Phe508del and previously eligible for Symkevi (Tezacaftor/Ivacaftor)
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)
- p.Phe508del heterozygous genotype: People with CF with 1 copy of p.Phe508del and not previously eligible for any CFTR modulator
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — MRI to study gut function and transit without the risk of exposure to ionising radiation.

SUMMARY:
An observational study of patients with cystic fibrosis (CF) starting treatment with Kaftrio (Elexacaftor / Tezacaftor / Ivacaftor) as part of routine clinical care, following EMA licensing (approved end of Aug 2020).

* Patients with CF who are p.Phe508del homozygotes will already be receiving the less effective CFTR modulator drug Symkevi (Tezacaftor / Ivacaftor) and will switch to KaftrioTM.
* Patients who are who are compound heterozygotes with at least 1 copy of p.Phe508del currently have access to no effective CFTR modulator and will be starting a CFTR modulator (Kaftrio) for the first time.

Participants attend a study visit before Kaftrio treatment commences, followed by visits at 12 and 24 weeks after starting treatment. At each visit they will be scanned before and after standardised meals in the morning and mid-day (11 scans in total over 6 hours). No intravenous contrast or bowel preparation will be used. Participants will complete questionnaires on gastrointestinal symptoms as well as providing stool and sputum samples for assessment of microbiome and stool for inflammatory mediators and pancreatic function (elastase).

**Following an extension, participants had a further visit at 76 weeks post starting Kaftrio, updated in detailed description**

DETAILED DESCRIPTION:
This is an observational study to observe the effects of Kaftrio (Elexacaftor / Tezacaftor / Ivacaftor) on the gut in people with CF.

Participants will attend 4 times, following an extension (pre-Kaftrio, at 12 weeks of Kaftrio at 24 weeks of Kaftrio and 76 weeks of Kaftrio) for MRI scanning at the Sir Peter Mansfield Imaging Centre, after an overnight fast. On this day, participants will be asked to withhold any medicines directly altering bowel habit such as laxatives. They will continue to take pancreatic enzyme replacement therapy and other medications for CF.

The Investigators will use the same MRI protocol as described in GIFT-CF (NCT03566550 and NCT04006873). Participants will have their first MRI scan fasted. After the first scan, they will eat a first standardised meal . They will then have 7 MRI scans at half hourly intervals and 3 MRI scans at hourly intervals. Participants will be given a second standardised meal after their ninth MRI scan. Each MRI scan will last approximately 15 minutes. After each MRI scan, participants will complete a validated gastrointestinal symptom questionnaire (Gastrointestinal Symptom Rating Scale). In between scans, participants will have access to an adjacent room with Wifi and television access.

They will also complete gut symptom questionnaires relating to the preceding 2 weeks and a 3 day food diary. They will also provide a sputum and stool sample.

Infection control requirements mean that only 1 participant will attend for MRI scanning per day. Extra COVID-19 precautions will also be taken throughout scan days.

***Please note, due to the timing of EMA approval for Kaftrio and ethics approval for the study granted on 21st Ocober 2020, the clinicaltrials.gov registration was created on 21st October 2020 and approved by the clinicaltrials.gov PRS team on 4th November 2020.***

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 60 years
* Capacity to consent, or to understand the requirements of the study where parental consent is needed.
* Confirmed diagnosis of CF, either by sweat test or genetic testing.
* Genotype homozygous p.Phe508del or compound heterozygous with at least 1 copy of p.Phe508del.
* Eligible for KaftrioTM (Elexacaftor / Tezacaftor / Ivacaftor) treatment but not yet commenced Kaftrio treatment as part of routine care.

Exclusion Criteria:

* Contra-indication to MRI scanning, such as embedded metal, pacemaker.
* FEV1 < 40% (% predicted using Global Lung Initiative values)
* Unable to stop medications directly prescribed to alter bowel habit, such as laxatives of anti-diarrhoeals, on the study day
* Previous resection of small bowel >20cm in length
* Intestinal stoma
* Diagnosis of inflammatory bowel disease or coeliac disease, confirmed by biopsy
* Gastrointestinal malignancy
* Unable to comply with dietary restrictions required for the study
* Pregnancy - tests are available at the SPMIC if participants are unsure
* Unable to speak or understand English

Ages: 12 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: All CF patients who receive care by Nottingham University Hospitals NHS Trust and are eligible for the study will be approached by their usual care team.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Difference in oro-caecal transit time (OCTT) in minutes at baseline and 24 weeks and baseline and 76 weeks | 4 days of scanning
  the time when the test meal is first detectable in the caecum

SECONDARY OUTCOMES:
Small bowel water content (SBWC) area under the curve (AUC), corrected for body surface area, measured in L.min/m^2 between 0 and 360 minutes at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of small bowel water representing secretions
Change in SBWC between 240 and 300 minutes (delta DTI) at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  These are small bowel water measurements before and after the second test meal
Colonic volume area under the curve (AUC), corrected for body surface area at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  volume of colon representing ease of chyme passage through colon
Stool calprotectin at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of gut inflammation
Stool and sputum microbiome at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of types of microbiome present in the stool and sputum
Stool elastase at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A marker of pancreatic exocrine function
Terminal ileum motility at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of motility at the terminal ileum using the GIQuant tool in arbitrary units
Abdominal symptoms as measured by the CFAbd-Score | 4 days of scanning
  A measure of gut symptoms over the preceding 2 weeks and during the study day, where a high score indicates more severe abdominal symptoms
Abdominal symptoms as measured by the PAC-SYM score | 4 days of scanning
  A measure of gut symptoms over the preceding 2 weeks and during the study day, where a high score indicates more severe abdominal symptoms
Abdominal symptoms as measured by 3 domains from the Gastrointestinal Symptoms Rating Scale (GSRS) | 4 days of scanning
  A measure of gut symptoms over the preceding 2 weeks and during the study day,, where a high score indicates more severe abdominal symptoms
Spirometry (FEV1) at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of lung function
Weight (kg) at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of body mass
Height (m) at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of growth

OTHER OUTCOMES:
T1 relaxation of ascending colon chyme at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  An approximate measure of water content in chyme present in the ascending colon
T2* of the terminal ileum | 4 days of scanning
  An approximate measure of gas bubbles in the terminal ileum
Terminal ileum diameter at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  A measure of the diameter of the terminal ileum in millimeters
Terminal ileum volume at baseline,12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  Volume of the terminal ileum
Colonic volume area under the curve, corrected for body surface area, of individual segments of the colon i.e. ascending, transverse, descending and rectosigmoid colon at baseline, 12 weeks, 24 weeks and 76 weeks | 4 days of scanning
  Volume of the ascending colon, transverse colon, descending colon and rectosigmoid colon representing of chyme/faeces passage through individual segments of the colon

CONTACTS AND LOCATIONS:
Overall Officials: Alan Smyth, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom